CLINICAL TRIAL: NCT04767373
Title: A Phase 2b/3 Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of MK-1654 in Healthy Pre-Term and Full-Term Infants
Brief Title: Efficacy and Safety of Clesrovimab (MK-1654) in Infants (MK-1654-004)
Acronym: CLEVER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1654-004; MK-1654-004 (Other: MSD); jRCT2051210019 (Registry Identifier: jRCT); PHRR210706-003684 (Registry Identifier: PHRR); 2022-500350-42-00 (Registry Identifier: EU CT); U1111-1275-5918 (Registry Identifier: UTN); 2020-002405-26 (EudraCT Number)
Record Dates: First submitted 2021-02-22; First posted 2021-02-23 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Syncytial Virus Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — MK-1654

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clesrovimab 105 mg (Experimental): Participants receive a single intramuscular (IM) administration of clesrovimab 105 mg on Day 1. An eligible subset of participants from RSV Season 1 will enter RSV season 2.
  Interventions: Biological: Clesrovimab
- Placebo (Placebo Comparator): Participants receive a single IM administration of placebo on Day 1. An eligible subset of participants from RSV Season 1 will enter RSV season 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Clesrovimab — Clesrovimab solution
  Other Names: MK-1654
  Arms: Clesrovimab 105 mg
Drug: Placebo — Placebo (0.9% sodium chloride [NaCL]) solution
  Arms: Placebo

SUMMARY:
The primary objectives of this phase 2b/3 double-blind, randomized, placebo-controlled study are to evaluate the efficacy and safety of clesrovimab in healthy pre-term and full-term infants. It is hypothesized that clesrovimab will reduce the incidence of respiratory syncytial virus (RSV)-associated medically attended lower respiratory infection (MALRI) from Days 1 through 150 postdose compared to placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Is a healthy male or female who is an early or moderate pre-term infant (≥29 to 34 weeks and 6 days gestational age) or a late pre-term or full-term infant (≥35 weeks gestational age)
* For the phase 2b cohort only: Has a chronological age >2 weeks of age up to 1 year and is entering their first respiratory syncytial virus (RSV) season at the time of obtaining documented informed consent.
* For the phase 3 cohort only: Has a chronological age from birth up to 1 year and is entering their first RSV season at the time of obtaining documented informed consent.
* For participants in South Korea only: Weighs ≥2 kg

Key Exclusion Criteria:

* Is recommended to receive palivizumab per local guidelines or professional society recommendations.
* Has known hypersensitivity to any component of clesrovimab
* Has a bleeding disorder contraindicating IM administration
* Has had a recent illness with rectal temperature ≥100.5°F (≥38.1°C) or axillary temperature ≥100.0°F (≥37.8°C) within 72 hours predose
* Has received any vaccine or monoclonal antibody for the prevention of RSV
* Is currently participating in or has participated in an interventional clinical study with an investigational compound or device at any time before first dose administration or while participating in this study

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3632 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (217):
- United States (51):
  - Southeastern Pediatric Associates, P.A. ( Site 0008), Dothan, Alabama
  - Northwest Arkansas Pediatric Clinic ( Site 0050), Fayetteville, Arkansas
  - Children's Clinic of Jonesboro, PA ( Site 0058), Jonesboro, Arkansas
  - Long Beach Memorial Medical Center ( Site 0014), Long Beach, California
  - Madera Family Medical Group ( Site 0046), Madera, California
  - Orange County Research Institute ( Site 0057), Ontario, California
  - Children's Hospital Colorado ( Site 0066), Aurora, Colorado
  - Optumcare Colorado Springs, LLC ( Site 0022), Colorado Springs, Colorado
  - Children's National Hospital ( Site 0076), Washington D.C., District of Columbia
  - MedStar Georgetown Pediatrics ( Site 0047), Washington D.C., District of Columbia
  - Next Phase Research Alliance, LLC ( Site 0071), Homestead, Florida
  - Acevedo Clinical Research Associates ( Site 0002), Miami, Florida
  - Tekton Research ( Site 0080), Chamblee, Georgia
  - Meridian Clinical Research, LLC ( Site 0083), Macon, Georgia
  - Clinical Research Prime ( Site 0075), Idaho Falls, Idaho
  - Saltzer Medical Group ( Site 0004), Nampa, Idaho
  - Cotton-O'Neil Clinical Research Center PediatricCare ( Site 0061), Topeka, Kansas
  - ACC Pediatric Research ( Site 0067), Haughton, Louisiana
  - Meridian Clinical Research, LLC ( Site 0082), Hastings, Nebraska
  - Midwest Children's Health Research Institute, LLC ( Site 0044), Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center ( Site 0031), Lebanon, New Hampshire
  - Rutgers University-Pediatric Clinical Research Center ( Site 0055), New Brunswick, New Jersey
  - Javara - Wake Forest Health Network - Ford, Simpson, Lively & Rice Pediatrics ( Site 0093), Winston-Salem, North Carolina
  - Senders Pediatrics ( Site 0062), Cleveland, Ohio
  - Ohio Pediatric Research Association ( Site 0063), Dayton, Ohio
  - CCP- Kid's Way ( Site 0017), Hermitage, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh - Primary Care Center - Oakland ( Site 0043), Pittsburgh, Pennsylvania
  - Coastal Pediatric Research ( Site 0013), Charleston, South Carolina
  - Tribe Clinical Research, LLC ( Site 0015), Greenville, South Carolina
  - Holston Medical Group ( Site 0040), Kingsport, Tennessee
  - Javara - Privia Medical Group North Texas - Frisco ( Site 0086), Frisco, Texas
  - University of Texas Medical Branch at Galveston ( Site 0059), Galveston, Texas
  - DM Clinical Research ( Site 0005), Houston, Texas
  - FMC Science - Lampasas ( Site 0011), Lampasas, Texas
  - DCOL Center for Clinical Research ( Site 0042), Longview, Texas
  - University Health System- San Antonio ( Site 0048), San Antonio, Texas
  - Private Practice - Dr. Etokhana ( Site 0089), San Antonio, Texas
  - Road Runner Research, Ltd ( Site 0049), San Antonio, Texas
  - Alliance for Multispecialty Research, LLC ( Site 0092), Kaysville, Utah
  - Wee Care Pediatrics ( Site 0077), Layton, Utah
  - Cottonwood Pediatrics ( Site 0032), Murray, Utah
  - Wee Care Pediatrics-Roy ( Site 0053), Roy, Utah
  - University of Utah School of Medicine ( Site 0006), Salt Lake City, Utah
  - Copperview Medical Center ( Site 0078), South Jordan, Utah
  - Wee Care Pediatrics ( Site 0065), Syracuse, Utah
  - Pediatric Research of Charlottesville, LLC ( Site 0073), Charlottesville, Virginia
  - MultiCare Rockwood Cheney Clinic ( Site 0068), Cheney, Washington
  - Multicare Health System Institute for Research and Innovation ( Site 0025), Spokane, Washington
  - Multicare Institute For Research And Innovation ( Site 0045), Tacoma, Washington
  - Marshall University School of Medicine and Medical Center ( Site 0064), Huntington, West Virginia
  - Marshfield Clinic ( Site 0054), Marshfield, Wisconsin
- Argentina (5):
  - Hospital Militar Central Cir Mayor Cosme Argerich ( Site 1001), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Clinica del Nino y la Madre ( Site 1005), Mar de La Plata, Buenos Aires
  - SANATORIO DEL SALVADOR-Pediatria ( Site 1008), Córdoba, Córdoba Province
  - SANATORIO MATER DEI ( Site 1010), Buenos Aires
  - Clinica Privada del Sol S.A ( Site 1013), Córdoba
- Belgium (5):
  - Universitair Ziekenhuis Antwerpen ( Site 2001), Edegem, Antwerpen
  - Centre Hospitalier Universitaire Saint Pierre (Bruxelles) ( Site 2003), Brussels, Bruxelles-Capitale, Region de
  - Cliniques Universitaires Saint-Luc ( Site 2005), Brussels, Bruxelles-Capitale, Region de
  - Cabinet Médical Demeulemeester ( Site 2002), Gozée, Wallonne, Region
  - AZ Delta ( Site 2004), Roeselare, West-Vlaanderen
- Canada (7):
  - University of Calgary - Alberta Children Hospital ( Site 0504), Calgary, Alberta
  - BC Women s Hospital and Health Centre ( Site 0506), Vancouver, British Columbia
  - Canadian Center for Vaccinology ( Site 0503), Halifax, Nova Scotia
  - Hamilton Medical Research Group ( Site 0509), Hamilton, Ontario
  - CHU Sainte Justine ( Site 0502), Montreal, Quebec
  - McGill University Health Centre - Vaccine Study Centre ( Site 0500), Pierrefonds, Quebec
  - CHU de Quebec Universite de Laval ( Site 0501), Québec, Quebec
- Chile (4):
  - Hospital La Florida ( Site 1104), Santiago, Region M. de Santiago
  - Hospital Roberto del Rio ( Site 1106), Santiago, Region M. de Santiago
  - Facultad Medicina Universidad de Chile ( Site 1105), Santiago, Region M. de Santiago
  - Hospital Padre Hurtado ( Site 1101), Santiago, Region M. de Santiago
- China (30):
  - Peking University Third Hospital ( Site 3339), Beijing, Beijing Municipality
  - The Children's Hospital of Chongqing Medical University ( Site 3333), Chongqing, Chongqing Municipality
  - Jiangjin District Central Hospital ( Site 3319), Chongqing, Chongqing Municipality
  - Xiamen Maternity and Child Health Care Hospital ( Site 3351), Xiamen, Fujian
  - Guangdong Provincial People's Hospital ( Site 3341), Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangzhou Medical University ( Site 3348), Guangzhou, Guangdong
  - Guangdong Maternity and Child Health Care Hospital ( Site 3340), Guangzhou, Guangdong
  - Liuzhou People's Hospital ( Site 3364), Liuchow, Guangxi
  - Hebei Petro China Central Hospital ( Site 3365), Langfang, Hebei
  - Fourth Hospital of Hebei Medical University ( Site 3366), Shijiazhuang, Hebei
  - Sanmenxia Central Hospital ( Site 3360), Sanmenxia, Henan
  - Wuhan Children's Hospital ( Site 3329), Wuhan, Hubei
  - Renmin Hospital of Wuhan University ( Site 3316), Wuhan, Hubei
  - Changde First People's Hospital ( Site 3311), Changde, Hunan
  - The Maternal and Child Health Hospital of Hunan Province ( Site 3334), Changsha, Hunan
  - Hunan Provincial People's Hospital ( Site 3355), Changsha, Hunan
  - Xiangya Hospital Central South University ( Site 3347), Changsha, Hunan
  - Hunan Shaoyang No.1 People's Hospital ( Site 3345), Shaoyang, Hunan
  - Zhongda Hospital Southeast University ( Site 3353), Nanjing, Jiangsu
  - Jiangxi Provincial Children's Hospital ( Site 3313), Nanchang, Jiangxi
  - The Third Hospital of Nanchang ( Site 3325), Nanchang, Jiangxi
  - Jiangxi Pingxiang People's Hospital ( Site 3312), Pingxiang, Jiangxi
  - Dalian Women and Children Medical Treatment Center(Hope Square Children's Branch Hospital) ( Site 33, Dalian, Liaoning
  - Children's Hospital of Fudan University ( Site 3361), Shanghai, Shanghai Municipality
  - Linfen Central Hospital ( Site 3368), Linfen, Shanxi
  - Linfen People's Hospital ( Site 3363), Linfen, Shanxi
  - Yuncheng Central Hospital - Eastern Hospital ( Site 3318), Yuncheng, Shanxi
  - Chengdu Women and Children Center Hospital ( Site 3332), Chengdu, Sichuan
  - The First People's Hospital of Hangzhou ( Site 3342), Hangzhou, Zhejiang
  - Ningbo Women and Children's Hospital ( Site 3314), Ningbo, Zhejiang
- Colombia (5):
  - Universidad Pontificia Bolivariana - Clinica Universitaria Bolivariana ( Site 1154), Medellín, Antioquia
  - Sociedad Medica de Rionegro SOMER S.A. ( Site 1157), Rionegro, Antioquia
  - Clinica de la Costa S.A.S. ( Site 1152), Barranquilla, Atlántico
  - Centro de Atención e Investigación Médica SAS - CAIMED CHIA ( Site 1155), Chía, Cundinamarca
  - Centro de Estudios en Infectologia Pediatrica SAS ( Site 1159), Cali, Valle del Cauca Department
- Denmark (4):
  - Regionshospitalet Herning ( Site 2105), Herning, Central Jutland
  - Aalborg Universitetshospital, Nord-Børne- og Ungeafdelingen ( Site 2100), Aalborg, North Denmark
  - Regionshospitalet Nordjylland ( Site 2102), Hjørring, North Denmark
  - Odense University Hospital ( Site 2107), Odense, Region Syddanmark
- Finland (10):
  - FVR, Kokkolan rokotetutkimusklinikka ( Site 2157), Kokkola, Keski-Pohjanmaa
  - FVR, Oulun rokotetutkimusklinikka ( Site 2158), Oulu, North Ostrobothnia
  - Tampereen yliopisto - Tampereen rokotetutkimusklinikka ( Site 2160), Tampere, Pirkanmaa
  - FVR, Porin rokotetutkimusklinikka ( Site 2156), Pori, Satakunta
  - FVR, Seinäjoen rokotetutkimusklinikka ( Site 2155), Seinäjoki, South Ostrobothnia
  - FVR, Turun rokotetutkimusklinikka ( Site 2151), Turku, Southwest Finland
  - FVR, Espoon rokotetutkimusklinikka ( Site 2152), Espoo, Uusimaa
  - FVR, Etelä-Helsingin rokotetutkimusklinikka ( Site 2159), Helsinki, Uusimaa
  - FVR, Itä-Helsingin rokotetutkimusklinikka ( Site 2153), Helsinki, Uusimaa
  - FVR, Järvenpään rokotetutkimusklinikka ( Site 2154), Jarvenpaa, Uusimaa
- France (3):
  - CHU Caen ( Site 2212), Caen, Calvados
  - Groupe Hospitalier Pellegrin ( Site 2218), Bordeaux, Gironde
  - Centre Hospitalier de Versailles ( Site 2206), Le Chesnay, Yvelines
- Israel (5):
  - Soroka Medical Center ( Site 2351), Beersheba
  - Soroka University Medical Center Ramot Family health center ( Site 2354), Beersheba
  - Rambam Medical Center ( Site 2352), Haifa
  - Soroka University Medical Center Rahat Family health center ( Site 2355), Rahat
  - Chaim Sheba Medical Center ( Site 2353), Ramat Gan
- Italy (5):
  - Policlinico Universitario Gemelli ( Site 2301), Rome, Roma
  - A.O.Universitaria Meyer ( Site 2306), Florence, Tuscany
  - Universita degli studi di Padova Patologia e TIN ( Site 2305), Padua, Veneto
  - A.O. Policlinico Consorziale di Bari ( Site 2309), Bari
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico ( Site 2310), Milan
- Japan (12):
  - Maebashi Red Cross Hospital ( Site 3057), Maebashi, Gunma
  - St. Marianna University School of Medicine Hospital ( Site 3060), Kawasaki, Kanagawa
  - JOHAS Yokohama Rosai Hospital ( Site 3058), Yokohama, Kanagawa
  - National Hospital Organization Beppu Medical Center ( Site 3063), Beppu, Oita Prefecture
  - Ageo Central General Hospital ( Site 3051), Ageo, Saitama
  - Tottori University Hospital ( Site 3053), Yonago, Tottori
  - Fukui Aiiku Hospital ( Site 3056), Fukui
  - Fukui-ken Saiseikai Hospital ( Site 3064), Fukui
  - Saitama City Hospital ( Site 3055), Saitama
  - Shizuoka City Shimizu Hospital ( Site 3061), Shizuoka
  - St.Luke's International Hospital ( Site 3062), Tokyo
  - Showa University Hospital ( Site 3059), Tokyo
- Malaysia (7):
  - Hospital Raja Perempuan Zainab II ( Site 3106), Kota Bharu, Kelantan
  - Hospital Seri Manjung ( Site 3103), Seri Manjung, Perak
  - Hospital Taiping ( Site 3108), Taiping, Perak
  - Hospital Pulau Pinang ( Site 3104), George Town, Pulau Pinang
  - Hospital Seberang Jaya ( Site 3107), Seberang Jaya, Pulau Pinang
  - Sabah Womens & Childrens Hospital ( Site 3102), Kota Kinabalu, Sabah
  - Hospital Sibu ( Site 3101), Sibu, Sarawak
- Mexico (4):
  - CAIMED Investigación en Salud S.A de C.V ( Site 1209), Mexico City, Mexico City
  - Centenario Hospital Miguel Hidalgo ( Site 1204), Aguascalientes
  - Hospital Angeles Lomas ( Site 1207), Huixquilucan
  - Instituto Nacional de Pediatria ( Site 1202), Mexico City
- Peru (4):
  - Clinica Peruano Americana S.A. ( Site 1253), Trujillo, La Libertad
  - Asociacion Civil Selva Amazonica ( Site 1255), Iquitos, Loreto
  - Hospital Nacional Docente Madre - Nino San Bartolome ( Site 1251), Lima
  - Instituto de Investigacion Nutricional - Anexo Huascar ( Site 1252), Lima
- Philippines (3):
  - University of the Philippines-Philippine General Hospital ( Site 3152), Manila, National Capital Region
  - Philippine Children s Medical Center ( Site 3154), Quezon City, National Capital Region
  - Far Eastern University - Nicanor Reyes Medical Foundation ( Site 3153), Quezon City, National Capital Region
- Poland (16):
  - Instytut Mikroekologii Sp. Z o.o. & Co. Sp. Komandytowa ( Site 2412), Poznan, Greater Poland Voivodeship
  - IN VIVO ( Site 2401), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne PROMED ( Site 2432), Krakow, Lesser Poland Voivodeship
  - Alergo-Med Specjalistyczna Przychodnia Lekarska SP ( Site 2403), Tarnów, Lesser Poland Voivodeship
  - Szpital im. sw. Jadwigi Slaskiej w Trzebnicy ( Site 2409), Trzebnica, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny-Klinika Pediatrii i Chorob Infekcyjnych ( Site 2440), Wroclaw, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Dzieciecy w Lublinie ( Site 2404), Lublin, Lublin Voivodeship
  - NZOZ Salmed ( Site 2433), Łęczna, Lublin Voivodeship
  - MTL Centrum Medyczne Puławska Społka zoo Sp K. ( Site 2426), Mazowieckie, Masovian Voivodeship
  - Szpital Kliniczny im Ks Anny Mazowieckiej ( Site 2435), Warsaw, Masovian Voivodeship
  - WIP Warsaw IBD Point Profesor Kierkus ( Site 2441), Warsaw, Masovian Voivodeship
  - Szpital Bielanski im. Ks. Jerzego Popiełuszki SPZOZ ( Site 2425), Warsaw, Masovian Voivodeship
  - Centrum Medyczne Pratia Warszawa ( Site 2438), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 2437), Gdansk, Pomeranian Voivodeship
  - Szpital Miejski w Tychach ( Site 2442), Tychy, Silesian Voivodeship
  - Gravita Diagnostyka i Leczenie Nieplodnosci ( Site 2423), Lodz, Łódź Voivodeship
- Romania (4):
  - Spitalul Clinic de Urgenta pentru Copii Brasov ( Site 2456), Brasov
  - Spitalul Clinic "Filantropia" Clinica Obstetrica-Ginecologie ( Site 2451), Bucharest
  - Spitalul Clinic Judetean De Urgenta Constanta ( Site 2458), Constanța
  - Spitalul Cinic de Obstretica si Ginecologie Cuza Voda ( Site 2452), Iași
- South Africa (7):
  - University Of The Orange Free State ( Site 2507), Bloemfontein, Free State
  - Baragwanath Hospital ( Site 2501), Johannesburg, Gauteng
  - Empilweni Services and Research Unit ( Site 2504), Johannesburg, Gauteng
  - Steve Biko Academic Hospital ( Site 2505), Pretoria, Gauteng
  - Enhancing Care Foundation-DICRS ( Site 2506), Durban, KwaZulu-Natal
  - Tygerberg Hospital ( Site 2503), Cape Town, Western Cape
  - MRC Unit on Child And Adolescent Health-Department of Paediatrics and child Health ( Site 2502), Cape Town, Western Cape
- South Korea (11):
  - The Catholic University of Korea, Incheon St. Mary's Hospital ( Site 3209), Bupyeong-gu, Incheon
  - Jeonbuk National University Hospital ( Site 3210), Jeonju, Jeonrabugdo
  - Korea University Ansan Hospital ( Site 3212), Ansan-si, Kyonggi-do
  - Hallym University Sacred Heart Hospital ( Site 3207), Anyang, Kyonggi-do
  - Seoul National University Bundang Hospital-Pediatrics ( Site 3204), Seongnam, Kyonggi-do
  - Pusan National University Hospital ( Site 3206), Busan, Pusan-Kwangyokshi
  - Chungang University Hospital ( Site 3211), Dongjak-gu, Seoul
  - Seoul National University Hospital ( Site 3203), Seoul
  - Severance Hospital Yonsei University Health System ( Site 3201), Seoul
  - Samsung Medical Center ( Site 3202), Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital ( Site 3208), Seoul
- Thailand (5):
  - Chulalongkorn University-Pediatrics ( Site 3252), Bangkok, Bangkok
  - Siriraj Hospital ( Site 3251), Bangkok, Bangkok
  - Srinagarind Hospital. Khon Kaen University ( Site 3253), Muang, Changwat Khon Kaen
  - Prince of Songkla University Faculty of Medicine ( Site 3255), Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital ( Site 3254), Chiang Mai
- Turkey (Türkiye) (5):
  - Cukurova Universitesi Tıp Fakultesi Balcalı Hastanesi ( Site 2555), Adana
  - Gazi Universitesi Saglık Arastırma ve Uygulama Merkezi ( Site 2552), Ankara
  - Ankara Universitesi Tip Fakultesi Cebeci Hastanesi ( Site 2551), Ankara
  - Ege University Medical Faculty ( Site 2553), Izmir
  - Erciyes University Medical Faculty-pediatric infection ( Site 2554), Kayseri
- United Kingdom (5):
  - UH Bristol Education Centre ( Site 2607), Bristol, Bristol, City of
  - St. Georges University Hospital NHS Foundation Trust ( Site 2601), London, London, City of
  - Royal Maternity Hospital ( Site 2602), Belfast, Northern Ireland
  - Oxford University Hospital NHS Foundation Trust ( Site 2604), Oxford, Oxfordshire
  - Alder Hey Childrens NHS Foundation Trust Hospital ( Site 2606), Liverpool

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Zar HJ, Simoes EAF, Madhi SA, Ramilo O, Senders SD, Shepard JS, Laoprasopwattana K, Piedrahita J, Novoa JM, Vargas SL, Dionne M, Jackowska T, Liu E, Ishihara Y, Ikeda K, Zhang Y, Railkar RA, Lutkiewicz J, Vora KA, Zang X, Maas BM, Lee AW, Guerra A, Sinha A; CLEVER (MK-1654-004) Study Group. Clesrovimab for Prevention of RSV Disease in Healthy Infants. N Engl J Med. 2025 Oct 2;393(13):1292-1303. doi: 10.1056/NEJMoa2502984. Epub 2025 Sep 17. PMID 40961446
- [Derived] Ginsburg AS, Srikantiah P. Respiratory syncytial virus: promising progress against a leading cause of pneumonia. Lancet Glob Health. 2021 Dec;9(12):e1644-e1645. doi: 10.1016/S2214-109X(21)00455-1. Epub 2021 Nov 11. No abstract available. PMID 34774184
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26484&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, participants received one dose of study treatment on Day 1 during RSV Season 1. Participants did not receive study treatment during RSV Season 2. Study disposition data were not collected separately for RSV season 1 and RSV Season 2.
Groups:
- Clesrovimab 105 mg: Participants received a single intramuscular (IM) administration of clesrovimab 105 mg on Day 1. An eligible subset of participants will be followed through RSV season 2.
- Placebo: Participants received a single IM administration of placebo on Day 1. An eligible subset of participants will be followed through RSV season 2.
Period: Overall Study
Arm/Group | Clesrovimab 105 mg | Placebo
Started | 2421 | 1211
Treated | 2411 | 1203
Safety Analysis Population (Per protocol, 3 participants who received study treatment were excluded from the safety analysis population due to protocol deviation.) | 2409 | 1202
Participants Who Entered RSV Season 2 | 1017 | 501
Completed | 2257 | 1126
Not Completed | 164 | 85
Not completed — Death | 6 | 3
Not completed — Lost to Follow-up | 67 | 35
Not completed — Physician Decision | 15 | 4
Not completed — Randomized By Mistake Without Study Treatment | 0 | 1
Not completed — Withdrawal By Parent/Guardian | 75 | 40
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Clesrovimab 105 mg | Placebo | Total
Number analyzed (Participants) | 2421 | 1211 | 3632
Age, Continuous [Mean (Standard Deviation); unit: Years] | 0.3 (0.2) | 0.3 (0.2) | 0.3 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1187 | 593 | 1780
  Male | 1234 | 618 | 1852
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 685 | 335 | 1020
  Not Hispanic or Latino | 1667 | 841 | 2508
  Unknown or Not Reported | 69 | 35 | 104
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 50 | 18 | 68
  Asian | 646 | 321 | 967
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 326 | 173 | 499
  White | 1085 | 553 | 1638
  More than one race | 304 | 139 | 443
  Unknown or Not Reported | 9 | 6 | 15
Region at randomization [Count of Participants; unit: Participants] — Region at randomization was categorized as the following: Northern hemisphere and Southern hemisphere.
  Participants
    Northern Hemisphere | 1657 | 818 | 2475
    Southern Hemisphere | 764 | 393 | 1157
Gestational Age [Count of Participants; unit: Participants] — Gestational age was categorized as the following: Early and Moderate Preterm Infant (≥29 to <35 weeks) Late Preterm and Full-term Infant (≥35 weeks)
  Participants
    Early and Moderate Preterm Infant (≥29 to <35 weeks) | 425 | 213 | 638
    Late Preterm and Full-term Infant (≥35 weeks) | 1996 | 998 | 2994
Age at randomization [Count of Participants; unit: Participants] — Age at randomization was categorized as <6 months and ≥6 months of age.
  Participants
    <6 months | 1927 | 964 | 2891
    ≥6 months | 494 | 247 | 741

OUTCOME MEASURES:

1. Primary Outcome: RSV Season 1: Number of Participants With Respiratory Syncytial Virus (RSV)-Associated Medically Attended Lower Respiratory Infection (MALRI)
Description: Outpatient and inpatient MALRI was defined as the presence of the following in a clinical setting: 1) cough or difficulty breathing; AND 2) 1 or more of wheezing, chest wall in-drawing/retraction, rales/crackles, hypoxemia, tachypnea, or dehydration due to respiratory symptoms; AND 3) RSV-positive reverse transcriptase polymerase chain reaction (RT-PCR) nasopharyngeal sample. Per protocol, the participants with outpatient and inpatient RSV-associated MALRI were reported together for RSV season 1 participants.
Time Frame: From Day 1 (postdose) to Day 150
Population: All randomized participants who received a dose of study treatment and were protocol compliant.
Measure: Count of Participants; unit: Participants
Groups:
- RSV Season 1: Clesrovimab 105 mg: Participants received a single intramuscular (IM) administration of clesrovimab 105 mg on Day 1.
- RSV Season 1: Placebo: Participants received a single IM administration of placebo on Day 1.
Arm/Group | RSV Season 1: Clesrovimab 105 mg | RSV Season 1: Placebo
Number analyzed (Participants) | 2398 | 1201
Participants | 60 | 74
Statistical Analysis 1: Comparison: RSV Season 1: Clesrovimab 105 mg vs RSV Season 1: Placebo; Test type: Other; p < 0.001, Exact method; One-sided p-value was estimated using an exact method; Efficacy estimate = 60.4, 95% CI 2-sided [44.1 to 71.9] — A modified Poisson regression with robust variance method was used to generate efficacy estimate (1- Relative Risk [RR]) & 95% confidence interval (CI). The model included region, gestational age, and age at randomization as covariates

2. Primary Outcome: RSV Season 1: Percentage of Participants With Solicited Injection-Site Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs included redness/erythema, swelling, and pain/tenderness. Per protocol, the percentage of RSV season 1 participants with solicited injection-site AEs were reported.
Time Frame: From Day 1 (postdose) to Day 5
Population: Safety analysis population included all randomized participants who received a dose of protocol specified study treatment. Per protocol, in the safety analysis population, participants with protocol deviation were excluded.
Measure: Number; unit: Percentage of participants
Arm/Group | RSV Season 1: Clesrovimab 105 mg | RSV Season 1: Placebo
Number analyzed (Participants) | 2409 | 1202
Percentage of participants | 11.4 | 11.7
Statistical Analysis 1: Comparison: RSV Season 1: Clesrovimab 105 mg vs RSV Season 1: Placebo; Test type: Other; Estimated Percentage Difference = -0.4, 95% CI 2-sided [-2.6 to 1.8] — Estimated percentage difference beteween Clesrovimab 105 mg arm and placebo arm and associated 95% CI were calculated based on the Miettinen & Nurminen method

3. Primary Outcome: RSV Season 1: Percentage of Participants With Fever
Description: Fever was defined as rectal temperature ≥102.2°F (≥39.0°C) or axillary temperature ≥101.7°F (≥38.7°C). Per protocol, the percentage of RSV season 1 participants with fever were reported.
Time Frame: From Day 1 (postdose) to Day 5
Population: Safety analysis population included all randomized participants who received a dose of protocol specified study treatment and had temperature data available. Per protocol, in the safety analysis population, participants with protocol deviation were excluded.
Measure: Number; unit: Percentage of participants
Arm/Group | RSV Season 1: Clesrovimab 105 mg | RSV Season 1: Placebo
Number analyzed (Participants) | 2408 | 1202
Percentage of participants | 0.5 | 1.2
Statistical Analysis 1: Comparison: RSV Season 1: Clesrovimab 105 mg vs RSV Season 1: Placebo; Test type: Other; Estimated Percentage Difference = -0.6, 95% CI 2-sided [-1.4 to -0.0] — Estimated percentage difference between Clesrovimab 105 mg arm and placebo arm and associated 95% CI were calculated based on the Miettinen & Nurminen method

4. Primary Outcome: RSV Season 1: Percentage of Participants With Solicited Systemic AEs
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited systemic AEs included irritability, somnolence/drowsiness, and appetite lost. Per protocol, the percentage of RSV season 1 participants with solicited systemic AEs were reported.
Time Frame: From Day 1 (postdose) to Day 5
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | RSV Season 1: Clesrovimab 105 mg | RSV Season 1: Placebo
Number analyzed (Participants) | 2409 | 1202
Percentage of participants | 30.1 | 31.2
Statistical Analysis 1: Comparison: RSV Season 1: Clesrovimab 105 mg vs RSV Season 1: Placebo; Test type: Other; Estimated Percentage Difference = -1.1, 95% CI 2-sided [-4.3 to 2.1] — [estimate comment as in outcome 3, analysis 1]

5. Primary Outcome: RSV Season 1: Percentage of Participants With Anaphylaxis/Hypersensitivity AE of Special Interest (AESI)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Anaphylaxis/Hypersensitivity AESI included anaphylaxis, angioedema, bronchospasm, drug hypersensitivity, dyspnea, hypersensitivity, dysphonia, and wheezing. Per protocol, the percentage of RSV season 1 participants with anaphylaxis/hypersensitivity AESI were reported.
Time Frame: From Day 1 (postdose) to Day 42
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | RSV Season 1: Clesrovimab 105 mg | RSV Season 1: Placebo
Number analyzed (Participants) | 2409 | 1202
Percentage of participants | 0.0 | 0.0
Statistical Analysis 1: Comparison: RSV Season 1: Clesrovimab 105 mg vs RSV Season 1: Placebo; Test type: Other; Estimated Percentage Difference = 0.0, 95% CI 2-sided [-0.3 to 0.2] — [estimate comment as in outcome 3, analysis 1]

6. Primary Outcome: RSV Season 1: Percentage of Participants With Rash AESI
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Rash AESI included acute generalized exanthematous pustulosis, drug eruption, drug reaction with eosinophilia and systemic symptoms, erythema multiforme, generalized rash of exfoliative nature, Stevens-Johnson syndrome, toxic epidermal necrolysis, and urticaria. Per protocol, the percentage of RSV season 1 participants with rash AESI were reported.
Time Frame: From Day 1 (postdose) to Day 42
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | RSV Season 1: Clesrovimab 105 mg | RSV Season 1: Placebo
Number analyzed (Participants) | 2409 | 1202
Percentage of participants | 0.5 | 0.3
Statistical Analysis 1: Comparison: RSV Season 1: Clesrovimab 105 mg vs RSV Season 1: Placebo; Test type: Other; Estimated Percentage Difference = 0.1, 95% CI 2-sided [-0.4 to 0.5] — [estimate comment as in outcome 3, analysis 1]

7. Primary Outcome: RSV Season 1: Percentage of Participants With ≥1 Nonserious AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Per protocol, the percentage of RSV season 1 participants with ≥1 nonserious AE were reported.
Time Frame: From Day 1 (postdose) to Day 42
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | RSV Season 1: Clesrovimab 105 mg | RSV Season 1: Placebo
Number analyzed (Participants) | 2409 | 1202
Percentage of participants | 74.8 | 75.5

8. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: An SAE was any untoward medical occurrence that results in death; is life-threatening; required inpatient hospitalization/prolongs existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or other important medical event. Per protocol, the percentage of participants in RSV season 1 and RSV season 2 with SAEs were reported.
Time Frame: RSV Season 1: Day 1 to Day 365, RSV Season 2: Day 366 to Day 515
Population: Safety analysis population which included all randomized participants who received a dose of protocol specified study treatment. For safety analysis population, participants with protocol deviation were excluded. Per protocol, a subset of participants from RSV season 1 entered RSV season 2 and SAEs were collected separately for RSV season 1 and RSV Season 2.
Measure: Number; unit: Percentage of participants
Groups:
- RSV Season 2: Clesrovimab 105 mg: A subset of participants from RSV season 1 entered RSV Season 2 per protocol. Participants received a single intramuscular (IM) administration of clesrovimab 105 mg on Day 1 during RSV Season 1.
- RSV Season 2: Placebo: A subset of participants from RSV season 1 entered RSV Season 2 per protocol. Participants received a single IM administration of placebo on Day 1 during RSV Season 1.
Arm/Group | RSV Season 1: Clesrovimab 105 mg | RSV Season 1: Placebo | RSV Season 2: Clesrovimab 105 mg | RSV Season 2: Placebo
Number analyzed (Participants) | 2409 | 1202 | 1017 | 501
Percentage of participants | 11.7 | 12.6 | 3.1 | 4.0

9. Secondary Outcome: RSV Season 1: Number of Participants With RSV-Associated Hospitalization
Description: RSV-associated hospitalization is defined as a hospital admission for respiratory illness and RSV-positive RT-PCR nasopharyngeal sample. Per protocol, the number of participants with RSV-associated hospitalization were reported for RSV season 1.
Time Frame: From Day 1 (postdose) to Day 150
Population: All randomized participants who received a dose of study treatment and were protocol compliant.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV Season 1: Clesrovimab 105 mg | RSV Season 1: Placebo
Number analyzed (Participants) | 2398 | 1201
Participants | 9 | 28
Statistical Analysis 1: Comparison: RSV Season 1: Clesrovimab 105 mg vs RSV Season 1: Placebo; Test type: Other; p < 0.001, Exact method — One-sided p-value was estimated using an exact method; Efficacy estimate = 84.2, 95% CI 2-sided [66.6 to 92.6] — A modified Poisson regression with robust variance method was used to generate efficacy estimate (1- RR) & 95% CI. The model included region, gestational age, and age at randomization as covariates

10. Secondary Outcome: RSV Season 1: Number of Participants With RSV-Associated MALRI
Description: Outpatient and inpatient MALRI was defined as the presence of the following in a clinical setting: 1) cough or difficulty breathing; AND 2) 1 or more of wheezing, chest wall in-drawing/retraction, rales/crackles, hypoxemia, tachypnea, or dehydration due to respiratory symptoms; AND 3) RSV-positive RT-PCR nasopharyngeal sample. Per protocol, participants with outpatient and inpatient RSV-associated MALRI were reported together for RSV season 1 participants.
Time Frame: From Day 1 (postdose) to Day 180
Population: All randomized participants who received a dose of study treatment and were protocol compliant.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV Season 1: Clesrovimab 105 mg | RSV Season 1: Placebo
Number analyzed (Participants) | 2398 | 1201
Participants | 64 | 77
Statistical Analysis 1: Comparison: RSV Season 1: Clesrovimab 105 mg vs RSV Season 1: Placebo; Test type: Other; Efficacy estimate = 59.5, 95% CI 2-sided [43.3 to 71.1] — [estimate comment as in outcome 9, analysis 1]

ADVERSE EVENTS:
Time Frame: RSV Season 1: Day 1 to Day 365, RSV Season 2: Day 366 to Day 515
Description: All-cause mortality was reported on all randomized participants. Serious and nonserious AEs were reported in safety analysis population. Per protocol, 3 participants were excluded from the safety analysis population due to protocol deviation. Per protocol, only all-cause mortality and SAEs were collected for RSV season 1 and RSV season 2 separately. No data for nonserious AEs were collected during RSV Season 2.
Arm/Group | RSV Season 1: Clesrovimab 105 mg | RSV Season 1: Placebo | RSV Season 2: Clesrovimab 105 mg | RSV Season 2: Placebo
All-Cause Mortality (participants affected / at risk) | 7/2421 | 3/1211 | 0/1017 | 0/501
Serious Adverse Events (participants affected / at risk) | 282/2409 | 151/1202 | 32/1017 | 20/501
Other Adverse Events (participants affected / at risk) | 1432/2409 | 724/1202 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV Season 1: Clesrovimab 105 mg (N=2409) | RSV Season 1: Placebo (N=1202) | RSV Season 2: Clesrovimab 105 mg (N=1017) | RSV Season 2: Placebo (N=501)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congenital vesicoureteric reflux (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinopathy of prematurity (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cricopharyngeal dysfunction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Sudden infant death syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Milk allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bacterial tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bronchiolitis (Infections and infestations) | 32 (33) | 19 (22) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 16 (17) | 7 (7) | 2 (2) | 0 (0)
Bronchitis mycoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bullous impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 6 (6) | 7 (7) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Coronavirus pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dysentery (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 20 (20) | 7 (7) | 3 (3) | 1 (1)
Gastroenteritis adenovirus (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HIV infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Herpangina (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Laryngitis viral (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 13 (15) | 4 (4) | 0 (0) | 2 (2)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metapneumovirus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metapneumovirus pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae viral bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Parasitic gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 43 (46) | 30 (33) | 2 (2) | 3 (4)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 6 (6) | 2 (2) | 1 (1) | 1 (1)
Pneumonia escherichia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 2 (2) | 8 (8) | 2 (3) | 0 (0)
Pneumonia viral (Infections and infestations) | 7 (7) | 1 (1) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 5 (5) | 13 (13) | 1 (1) | 2 (2)
Respiratory syncytial virus infection (Infections and infestations) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 4 (4) | 4 (4) | 0 (0) | 2 (2)
Rhinolaryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Salmonella bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 12 (14) | 4 (4) | 0 (0) | 0 (0)
Varicella zoster pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Exposure to SARS-CoV-2 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeding disorder (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 10 (14) | 3 (3) | 2 (2) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motor developmental delay (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural effusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autism spectrum disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 2 (3) | 0 (0)
Brief resolved unexplained event (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Childhood asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibrinous bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cyanosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV Season 1: Clesrovimab 105 mg (N=2409) | RSV Season 1: Placebo (N=1202) | RSV Season 2: Clesrovimab 105 mg (N=0) | RSV Season 2: Placebo (N=0)
Diarrhoea (Gastrointestinal disorders) | 139 (155) | 77 (91) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 156 (159) | 96 (97) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 139 (158) | 78 (89) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 351 (415) | 189 (212) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 215 (253) | 108 (123) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 161 (176) | 93 (106) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 347 (393) | 199 (231) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 582 (789) | 303 (417) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 201 (254) | 93 (133) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 205 (256) | 98 (129) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 170 (220) | 72 (91) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may be published or presented at scientific meetings. The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Any information identified by the Sponsor as confidential must be deleted prior to submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT04767373/Prot_SAP_000.pdf